CLINICAL TRIAL: NCT01550341
Title: HIV, Buprenorphine, and the Criminal Justice System
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: George Mason University (Other); Howard University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011007631; R01DA030768 (NIH)
Record Dates: First submitted 2011-06-21; First posted 2012-03-12 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Opiate Addiction; Drug Dependence
Keywords: HIV; AIDS; Opiate Addiction; Drug Dependence; Buprenorphine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Active Comparator)
  Interventions: Drug: Buprenorphine/naloxone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Buprenorphine/naloxone — 2/0.5, 8/2 sublingual tabs; dosage based on medical assessment; medications taken once per day for 12 months duration.
  Other Names: Suboxone
  Arms: Buprenorphine
Drug: Placebo Oral Tablet — 2/0.5, 8/2 sublingual tabs; dosage based on medical assessment; medications taken once per day for 12 months duration.
  Arms: Placebo

SUMMARY:
The aims of STRIDE were changed as of July, 2014. The revised project, called STRIDE2, has a longitudinal, non-randomized, observational study design. The population under study consists of individuals living with HIV who are dependent on opioids.

DETAILED DESCRIPTION:
Presented in the results section are the summary of outcomes from the STRIDE RCT that were collected prior to the change in study design. The STRIDE study became STRIDE2 (NCT03583138). Those individuals originally enrolled in the STRIDE RCT will be followed for 12 months.

STRIDE2 will assist in identifying and monitoring individuals' HIV risk behaviors and provide resources to seek treatment for their HIV care and substance use. The goal of STRIDE2 is to examine if there are differences in HIV, drug use, and other outcomes between individuals receiving treatment versus individuals actively using, not actively using and not in treatment, and individuals on Methadone, Suboxone, or in some other treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Age ≥18 yrs
* Meets DSM-IV criteria for opioid dependence
* Has medical entitlements in DC
* Able to provide informed consent
* Able to communicate in English or Spanish

Exclusion Criteria:

* Being prescribed an opiate medication for a chronic pain condition or expressing the need to be placed on chronic pain medical conditions for a documented pain condition
* Currently receiving methadone dosing of over 30 mg per day and uninterested in changing to buprenorphine
* AST and ALT >5x the upper limit of normal (AST≥175, ALT≥195)
* Pregnant or unwilling to use contraception (including OCPs, patch, Depo-Provera, condoms, etc.)
* Breastfeeding or unwilling to stop breastfeeding
* Subject is part of another pharmacological research study
* Liver dysfunction (acute hepatitis, liver failure or hepatic dysfunction)
* Suicidal ideation
* Hypersensitivity to buprenorphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University School of Medicine/AIDS Program; Faye Taxman, PhD, Principal Investigator — George Mason University; William Lawson, MD, Principal Investigator — Howard University
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine | Placebo
Started | 32 | 18
Completed | 32 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Placebo | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 17 | 49
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.29 (6.54) | 55.59 (5.26) | 52.81 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 23 | 13 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 18 | 50

OUTCOME MEASURES:

1. Primary Outcome: CD4 Count Absolute
Description: CD4 Count Absolute
Time Frame: Baseline
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 31 | 13
cells/uL | 486.15 (308.34) | 403.92 (233.89)

2. Primary Outcome: CD4 Count Absolute
Description: CD4 Count Absolute
Time Frame: 6 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 31 | 18
cells/uL | 455.52 (289.74) | 551.23 (82.12)

3. Primary Outcome: CD4 Count Absolute
Description: CD4 Count
Time Frame: 12 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 31 | 18
cells/uL | 490.25 (298.65) | 492.33 (260.43)

4. Primary Outcome: CD4 Percent
Description: CD4 Percent
Time Frame: Baseline
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: CD4 Percent
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 31 | 13
CD4 Percent | 23.36 (8.56) | 25.7 (12.38)

5. Primary Outcome: CD4 Percent
Description: CD4 Percent
Time Frame: 6 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: CD4 Percent
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 31 | 13
CD4 Percent | 21.33 (1.88) | 28.56 (12.1)

6. Primary Outcome: CD4 Percent
Description: CD4 Percent
Time Frame: 12 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: CD4 Percent
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
CD4 Percent | 22.14 (9.6) | 27.95 (12.14)

7. Primary Outcome: Viral Load
Description: Viral Load
Time Frame: Baseline
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
IU/mL | 1465.00 (551.17) | 896.50 (1569.7)

8. Primary Outcome: Viral Load
Description: Viral Load
Time Frame: 6 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
IU/mL | 9269.04 (4778.9) | 7891.08 (26598.95)

9. Primary Outcome: Viral Load
Description: Viral Load
Time Frame: 12 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
IU/mL | 8122.10 (18268.77) | 19425.71 (51342.69)

10. Primary Outcome: Log Viral Load
Description: Log Viral Load
Time Frame: Baseline
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: log(IU/mL)
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
log(IU/mL) | 2.12 (1.02) | 2.00 (.97)

11. Primary Outcome: Log Viral Load
Description: Log Viral Load
Time Frame: 6 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: log(IU/mL)
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
log(IU/mL) | 2.22 (1.35) | 1.79 (1.11)

12. Primary Outcome: Log Viral Load
Description: Log Viral Load
Time Frame: 12 Months
Population: Participants with complete lab results.
Measure: Mean (Standard Deviation); unit: log(IU/mL)
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 32 | 18
log(IU/mL) | 2.40 (1.33) | 1.84 (1.44)

13. Secondary Outcome: Improved Opioid Treatment Outcomes
Description: Monitor relapse to opioid use, retention on Buprenorphine or placebo, percent days using opioids, lower addiction severity, lower craving, between baseline and subsequent follow-up visits. Monitor urine toxicology screens on every visit for approximately one year.
Time Frame: baseline, 3 months, 9 months, 12 months
Population: This outcome was not collected and analyzed due to the change in study design (see study description).
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Improved Criminal Justice Outcomes
Description: Measure change in time to reincarceration,number of days reincarcerated, and crime days, between baseline and each monthly follow-up visit.
Time Frame: baseline, wk 4, 9, 13, 18, 22, 27, 31, 36, 40, 45, 49, 52
Population: These data were never collected and summarized due to the change in study design (see study description).
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 0 | 00000

ADVERSE EVENTS:
Arm/Group | Buprenorphine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/18
Other Adverse Events (participants affected / at risk) | 0/32 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No